CLINICAL TRIAL: NCT05515250
Title: Neuromodulation With Percutaneous Electrical Nerve Field Stimulation for Children With Cystic Fibrosis Experiencing Chronic Abdominal Pain
Brief Title: Neuromodulation for Children With Cystic Fibrosis Experiencing Chronic Abdominal Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inadequate enrollment. Found only one participant over 1 year as opposed to anticipated over 15 patients. Inadequate research funding and staff support also added to this decision.
Sponsor: St. Louis University (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Dhiren Patel, MD, MBBS, MD Associate Professor of Pediatrics, Medical Director of Neurogastroenterology and Motility, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31972
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cystic Fibrosis; Irritable Bowel Syndrome; Chronic Pain
MeSH Terms: conditions — Cystic Fibrosis; Irritable Bowel Syndrome; Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patient open label intervention arm (Other)
  Interventions: Device: Use of neurostimulation device

INTERVENTIONS:
Device: Use of neurostimulation device — In humans, abdominal pain is modulated by the vagus nerve. Stimulation of the vagus nerve has been suggested to reduce visceral sensitivity and abdominal pain. IB-stim is the Percutaneous Electrical Nerve Field Stimulation (PENS) device. It is a non-invasive, outpatient therapy. PENFS has been shown to be efficacious in pediatric patients with abdominal pain.

SUMMARY:
Chronic abdominal pain is extremely common in individuals with Cystic Fibrosis (CF). Therapy for chronic abdominal pain is very limited and generally consists of osmotic laxatives or drugs that are used to treat irritable bowel syndrome (IBS), most of which are off-label and not proven to be effective for CF patients. Abdominal pain negatively impacts the quality of life (QOL). With the development of novel therapies for CF, life expectancy has significantly increased. There is, therefore, a critical need to identify treatment pathways for chronic abdominal pain in children with CF.

In humans, abdominal pain is modulated by the vagus nerve. Stimulation of the vagus nerve has been suggested to reduce visceral sensitivity and abdominal pain. IB-stim is the Percutaneous Electrical Nerve Field Stimulation (PENS) device. It is a non-invasive, outpatient therapy. PENFS has been shown to be efficacious in pediatric patients with abdominal pain. The FDA has cleared and classified this device as class II, suggesting minimal to moderate risk.

There is increasing evidence of intestinal inflammation in patients with CF, which could help explain the GI symptoms and differentiate from IBS. Studies have reported increased inflammation in the intestines using fecal calprotectin.

With the implementation of this study, investigators hypothesize that the IB -Stim device will reduce their overall GI inflammation and abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking and willing to consent and follow the study protocol
* Children with CF aged 11-17 years at the time of enrollment. All races, ethnic groups and both sexes will be included. Patient turning 18 years after enrollment in the study will continue in study and complete remaining study visits.
* Minimum of 2 days of abdominal pain/week for a duration of two months or greater prior to starting the study
* Average weekly abdominal pain score of at least 3 for the previous 2 weeks prior to entering the study (on a 0-10-point rating scale).
* Abdominal pain is not explained by any major organic etiology and comprehensive work up failed to identify any single cause for patients' symptoms

EXCLUSION CRITERIA:

* Patients age of 18 years and over, or less than 11 years at the time of enrollment
* Patients who cannot provide informed consent or do not speak English
* Patients with abdominal pain that can be explained clinically by other GI diagnoses other than CF per study doctor's judgement
* History of cranial nerve or major abdominal surgeries in last 6 months
* Patients with underlying neurologic conditions, including history of ongoing seizures or traumatic brain injury within last 6 months
* Patients with dermatologic conditions affecting the ears (i.e. psoriasis), or with cuts or abrasions to the external ear that would interfere with electrode placement
* Patients with hemophilia or other bleeding disorders
* Patients with any implanted electromagnetic device
* Inability to comply with study protocol and follow up, per study doctor's judgement.
* Pregnant females, females who are breastfeeding or who believe they may wish to become pregnant during the course of the study
* Males and females of reproductive potential who are unwilling to use effective measures (chosen in consultation with their health care provider) to avoid becoming pregnant.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Unsure about the number of participants and their willingness to allow us to share the data.

REFERENCES:
- [Background] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label: Only treatment Arm.
Period: Overall Study
Arm/Group | Open Label
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patient Open Label Intervention Arm
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: IBS Severity Scoring System-Change Between Baseline and Week 8 is Reported.
Description: IBS-SSS is a tool for assessing IBS. Please refer to the following for further understanding of this tool. It records Part 1- Severity Score( 0-500 where 0 is no symptom and 500 is the severe symptoms) and Part 2 ' Other IBS Data' under which includes bowel habits, consistency of bowel movements, red flag symptoms, site of pain and absence from work due to IBS. We cannot use part 2 because it does not have assigned scoring system and as such not suitable for patients with CF due to know genetic mutation in CF causing many similar symptoms of IBS. It has nine stem q: five questions ( in Part 1) have scores of between 0 and 100 for each question, based on visual analogue scales, each minimum of 0 to max of 100.We report combined sub score at baseline and week 8. A score below 75 is seen in healthy people or in remission of IBS, 75-175 indicates mild disease, 175-300 moderate disease and over 300 severe. The score is interpreted as an absolute change from the baseline and at week 8.
Time Frame: baseline and 8 weeks
Measure: Number; unit: score on a scale
Arm/Group | Patient Open Label Intervention Arm
Number analyzed (Participants) | 1
score on a scale
  IBS Severity Scoring System at baseline | 50
  IBS Severity Scoring System at week 8 | 25

2. Primary Outcome: CFQ-R and PedsQL Gastrointestinal Scale Score in Response to IB-Stim Treatment- Baseline and Week 8 Reported
Description: Name of categories/domains CFQ-R:
  9 Quality of life domains: Physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions.
  3 symptom scales: Weight, respiratory, and digestion. Scaling of items: 5 distinct 4-point Likert scales (e.g., always/often/ sometime/never)
  Scoring: Range from 0 to 100, with higher scores indicating better health.
  PedsQL consists of 74 items comprising 14 dimensions Likert scale from 0 to 4.Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0.Total Score: Sum of all the items over the number of items answered on all the Scales. PedsQL scoring interpretation: In general, the higher scores indicating better health for this measure.
  Baseline and week 8 reported
Time Frame: baseline and 8 weeks
Measure: Number; unit: score on a scale
Groups:
- Patient Open Label Intervention Arm: We report the following group in response to IB stim treatment:
  CFQ-R - Baseline CFQ-R- Week 8 PedsQL Gastrointestinal Scale Score- Baseline Peds QL Gastrointestinal Scale Score- week 8
Arm/Group | Patient Open Label Intervention Arm
Number analyzed (Participants) | 1
score on a scale
  CFQ-R score at baseline | 75
  PedsQL- Gastrointestinal Module score at baseline | 78
  CFQ-R score at week 8 | 70
  PedsQL- Gastrointestinal Module score at week 8 | 73

3. Primary Outcome: Reduction in Stool Calprotectin Inflammatory Markers in Response to IB-Stim-change Between Two Time Point is Reported.
Description: Investigators hypothesize that at 4 weeks following PENFS treatment initiation, there will be a reduction in stool calprotectin to baseline. The higher the value, worse the disease. The value above 200 ug/mg is considered to be suggestive of significant inflammation in the gut.
Time Frame: Baseline and week 4
Measure: Number; unit: μg/mg
Arm/Group | Patient Open Label Intervention Arm
Number analyzed (Participants) | 1
μg/mg
  Baseline | 36
  Week 4 | 30

ADVERSE EVENTS:
Time Frame: 2 month and 10 days
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Main plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT05515250/Prot_SAP_001.pdf